CLINICAL TRIAL: NCT04650035
Title: The Impact of COVID-19 on Surgical Practice in Jordan During the Second Outbreak : A Survey
Brief Title: The Impact of COVID-19 on Surgical Practice in Jordan During the Second Outbreak
Status: Completed | Type: Observational
Sponsor: Yarmouk University (Other)
Responsible Party: Principal Investigator, Raed M Ennab, Assistant Professor, Yarmouk University
Other Study IDs: The Impact of COVID-19 Jordan
Record Dates: First submitted 2020-12-01; First posted 2020-12-02 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: COVID-19 is an acute respiratory pandemic with no available effective antiviral treatment or widely available effective vaccine. Surgical practice has faced widespread problems due to the pandemic including viral transmission risk and cross-infection, staffing problems, prioritizations of surgical procedures and lack of beds due to occupancy of hospitals and ICU beds with COVID-19 patients; Methods: A survey was conducted between October 31 to November 4, 2020, through google forms. The questionnaire involved 16 questions sent to consultants and specialists of all general and special surgical specialties and subspecialties in Jordan;

DETAILED DESCRIPTION:
A survey was conducted between October 31 and November 4, 2020. The questionnaire was made through google forms, and a consent was taken from the Jordan medical association to send the link to surgeons in Jordan through the social media and the official WhatsApp groups. The survey was introduced with the invitation to participate of surgeons of all general and special surgical specialties and subspecialties. The aim of the survey was mentioned in the introduction which was to evaluate the impact of COVID-19 on surgical practice in Jordan during the second outbreak of COVID-19, and it was explained that the aim of the survey was for research purposes only and that it was totally anonymous with privacy preserved, and no identifying information required. Also, it was noted that we have added spaces for written views and recommendations.

The questionnaire involved 16 questions of the multiple-choice, the dropdown, the multiple check, and the short answer questions. The first 2 questions were about the specialty and the place of work whether it was the ministry of health, the royal medical services, the university hospitals, or the non-governmental organizations. The 3rd and 4th questions were about the hospital where the participant works whether it admits COVID-19 patients and/or ordinary patients. The Questions from the 5th to the 8th were about the volume of work in terms of the number of elective and emergency surgeries during the month of October 2020 in comparison to the average monthly rate during the year 2019. The questions from the 9th to the 15th were about the problems that might have been faced in managing elective and emergency cases during the month of October 2020 in relation to COVID-19. The last question was a multiple checkbox question with an added space for giving the possible recommendations to manage the situation.

ELIGIBILITY:
Inclusion Criteria:

* Consultants and specialists of all general and special surgical specialties and subspecialties in Jordan

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consultants and specialists of all general and special surgical specialties and subspecialties in Jordan
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Number of surgical operations performed whether elective or emergency | October 2020
  difference between the monthly rate of operations during 2019 and the month of October 2020.

CONTACTS AND LOCATIONS:
Overall Officials: Raed M Ennab, Study Director — Department of Clinical Sciences, Faculty Of Medicine, Yarmouk University
Locations (1):
- Yarmouk University, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo YR, Cao QD, Hong ZS, Tan YY, Chen SD, Jin HJ, Tan KS, Wang DY, Yan Y. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak - an update on the status. Mil Med Res. 2020 Mar 13;7(1):11. doi: 10.1186/s40779-020-00240-0. PMID 32169119
- [Background] Lam S, Lombardi A, Ouanounou A. COVID-19: A review of the proposed pharmacological treatments. Eur J Pharmacol. 2020 Nov 5;886:173451. doi: 10.1016/j.ejphar.2020.173451. Epub 2020 Aug 6. PMID 32768505
- [Background] Al-Jabir A, Kerwan A, Nicola M, Alsafi Z, Khan M, Sohrabi C, O'Neill N, Iosifidis C, Griffin M, Mathew G, Agha R. Impact of the Coronavirus (COVID-19) pandemic on surgical practice - Part 1. Int J Surg. 2020 Jul;79:168-179. doi: 10.1016/j.ijsu.2020.05.022. Epub 2020 May 12. PMID 32407799
- [Background] Coccolini F, Perrone G, Chiarugi M, Di Marzo F, Ansaloni L, Scandroglio I, Marini P, Zago M, De Paolis P, Forfori F, Agresta F, Puzziello A, D'Ugo D, Bignami E, Bellini V, Vitali P, Petrini F, Pifferi B, Corradi F, Tarasconi A, Pattonieri V, Bonati E, Tritapepe L, Agnoletti V, Corbella D, Sartelli M, Catena F. Surgery in COVID-19 patients: operational directives. World J Emerg Surg. 2020 Apr 7;15(1):25. doi: 10.1186/s13017-020-00307-2. PMID 32264898
- [Background] Russell FM, Greenwood B. Who should be prioritised for COVID-19 vaccination? Hum Vaccin Immunother. 2021 May 4;17(5):1317-1321. doi: 10.1080/21645515.2020.1827882. Epub 2020 Nov 3. PMID 33141000
- See also: Department of Statistics Jordan. Population Count. (2020). — http://dosweb.dos.gov.jo
- See also: Prime Ministry of Jordan. Official Reports. (2020). — http://www.pm.gov.jo/
- See also: Jordanian Ministry of Health. COVID-19 in Jordan. (2020). — https://corona.moh.gov.jo/ar
- See also: The American Board of Surgery official website, COVID-19 Guidelines and Resources — https://www.absurgery.org/default.jsp?covid19_resources